CLINICAL TRIAL: NCT02005991
Title: A Phase 1, Open-Label Study To Evaluate 5-HT2a Receptor Occupancy As Measured By Positron Emission Tomography (PET) With Ligand [11C]MDL100907 Following Single Oral Dose Administration Of PP-05212377 (SAM-760) In Healthy Subjects
Brief Title: A Study To Examine The Distribution Of PF-05212377 In The Brain Of Healthy Volunteer Subjects Using Positron Emission Tomography And A Radioactive Tracer Following Oral Administration Of One Dose Of PF-05212377
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: B2081015
Record Dates: First submitted 2013-11-05; First posted 2013-12-09 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-04

CONDITIONS: Healthy
Keywords: PF-05212377; phase 1; open-label; 5-HT2a receptor occupancy; positron emission tomography; healthy subjects; brain; cortex; alzheimers disease
MeSH Terms: conditions — Alzheimer Disease | interventions — SAM-760

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PF-05212377 70 mg (Experimental)
  Interventions: Drug: PF-05212377
- PF-05212377 20 mg (Experimental)
  Interventions: Drug: PF-05212377
- PF-05212377 10 mg (Experimental)
  Interventions: Drug: PF-05212377

INTERVENTIONS:
Drug: PF-05212377 — Single, oral dose administration of 70 mg PF-0521377 using a capsule formulation.
  Arms: PF-05212377 70 mg
Drug: PF-05212377 — Single, oral dose administration of 20 mg PF-0521377 using a capsule formulation. This dose is an estimate. The exact dose for Arm 2 will be based on the results from Arm 1.
  Arms: PF-05212377 20 mg
Drug: PF-05212377 — Single, oral dose administration of 10 mg PF-0521377 using a capsule formulation. This dose is an estimate. The exact dose for Arm 2 will be based on the results from Arms 1 and 2.
  Arms: PF-05212377 10 mg

SUMMARY:
This study will see how PF-05212377, an experimental drug to treat symptoms from Alzheimer's Disease, distributes in the brain after one dose of PF-05212377 is administered orally to healthy volunteer subjects. The study will also evaluate the safety and tolerability of PF-05212377 in these subjects and will measure the level of PF-05212377 in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Males and females must be at least 18 years of age and no older than 55 years of age with a Body Mass Index (BMI) must be between 17.5 and 30.5.
* Subjects must sign a consent form and comply with all scheduled visits, treatment plan, lab tests and other study procedures.

Exclusion Criteria:

* Females must not be pregnant, breastfeeding, or able to have children.
* Subjects must not have a severe acute or chronic medical or psychiatric condition history or evidence of blood, kidney, glandular, lung, stomach, intestine, heart, blood vessel, liver, psychiatric, nerve, or allergic problems (including drug allergies), except mild seasonal allergies.
* Subjects must not drink alcohol excessively or take illicit drugs.
* Male subjects use condoms to prevent the potential transfer of drug through the semen to their partner beginning with the dose of study drug and use a highly effective method of birth control with any partner(s) of childbearing potential through 28 days after the last dose.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2013-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
5-HT2a receptor occupancy of PF-05212377 in the frontal cortex using PET | Days 1 and 2
Plasma PF-05212377 exposure associated with PF-05212377 5-HT2a receptor occupancy | Days 1 and 2

SECONDARY OUTCOMES:
5-HT2a receptor occupancy of PF-05212377 in other cortical regions | Day 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2081015&StudyName=A%20Study%20To%20Examine%20The%20Distribution%20Of%20PF-05212377%20In%20The%20Brain%20Of%20Healthy%20Volunteer%20Subjects%20Using%20Positron%20Emission%20Tomography%20And%20A